CLINICAL TRIAL: NCT05410028
Title: New Serum Biomarkers for Monitoring Early Diagnosis of Ovarian Cancer Recurrence Via Analysis of Immunoinflammation-related Protein Complexes in Blood
Brief Title: New Serum Biomarkers for Monitoring Early Diagnosis of Ovarian Cancer Recurrence
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PUMCH-OC2
Record Dates: First submitted 2022-06-04; First posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-03

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1 mL of serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention in clinical treatment — No intervention in clinical treatment

SUMMARY:
In this study, mass spectrometry was used to analyze immune inflammation-related protein complexes, post-translational modified glycopeptide omics and tumor-related metabolomics in serum, respectively, in order to find potential metabolic small molecule biomarkers or marker profiles that can be used for early diagnosis of cancer recurrence.

DETAILED DESCRIPTION:
Time cohort study: patients with confirmed ovarian epithelial cancer at different time cutoff points before treatment, after surgery, during chemotherapy, and after chemotherapy, until clinically confirmed patients relapse. At least 50 patients are expected to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Female
* A diagnosed patient with epithelial ovarian cancer
* Age ≤ 70

Exclusion Criteria:

* Male
* Suffering from other malignant tumors
* Non-compliant patient
* Age above 70

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Before treatment, after surgery, during chemotherapy, and after chemotherapy, patients with confirmed ovarian epithelial cancer had different time cutoff points until clinically confirmed patients recurred.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-03-03 (Actual); Primary Completion 2024-03-03 (Estimated); Study Completion 2026-03-03 (Estimated)

PRIMARY OUTCOMES:
Immune Inflammation-Related Protein Complexes | 2 years
  The change of immune inflammation-related protein complexes

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No